CLINICAL TRIAL: NCT03870867
Title: Intracranial Bleeding and Emergency Physician CT Scanning in Seniors Who Have Fallen
Brief Title: The Emergency Department Falls Study
Acronym: FALLS
Status: Completed | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: 467
Record Dates: First submitted 2018-04-06; First posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Fall; Head Injury Trauma; Intracranial Hemorrhages
Keywords: seniors; falls; imaging; emergency department; CT head; intracranial hemorrhages
MeSH Terms: conditions — Intracranial Hemorrhages; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Seniors who have fallen: Emergency department patients over the age of 65 who present to the emergency department after a fall.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This is a pilot study to evaluate clinical predictors of intracranial bleeding in elderly patients who present to the emergency department (ED) after a fall. The aim is to assess feasibility and rate of patient recruitment, patient follow up, and to establish a point estimate for the incidence of intracranial bleeding in the investigator's population.

Currently there are no guidelines for ED physicians to assess the pretest probability of intracranial bleed in these patients, and no safe way to exclude a bleed without CT.

DETAILED DESCRIPTION:
Seniors account for 15% of the Canadian population. The proportion will greatly increase over the next few years. Elderly people attend the ED more often than younger people, and they often come to the ED after a fall at home or outside. Falling is associated with head injuries, which cause half of all the deaths from falling.

Head injuries are diagnosed with CT scans. In the ED, it can be difficult for the physician to know when to perform a CT scan of the head. It can be hard to know if the elderly person hit their head, and often times, people with bleeding in the head can have a normal examination. The Investigators think that the overall risk of bleeding in the head in elderly who fall is between 3 and 10%. If emergency physicians scanned every senior who fell, only a few would show bleeding, the scanning department would be overwhelmed, there would be increased costs for the hospital and longer delays for patients. It is important for physicians to diagnose a serious head injury as there are lifesaving treatments that can be given.

The Investigators plan to develop a decision rule for emergency physicians that would inform them which patients should have a CT scan of the head and which patients can have a serious head injury safely ruled out without a CT.

The Investigators propose to identify and recruit patients over the age of 65 who come to the Hamilton General or Juravinski Emergency departments after falling. Patients and their caregivers will be consented for a telephone follow-up call after 6 weeks. Data collected will include patient characteristics, general health, and blood test results which might be predictors of a serious head injury.

The Investigators will develop a tool to help emergency physicians to order a CT scan on the right patients.

ELIGIBILITY:
Inclusion Criteria:

* 65+ years
* Presenting to the emergency department with fall on level ground, from a bed, from a chair, from the toilet seat or down steps 1 or 2 steps, within the last 48 hours

Exclusion Criteria:

* Non-English speaking without an an adequate interpreter
* Falls with an other mechanism of injury
* Falls > 48 hours before presentation

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients over the age of 65 who present to the emergency departments of the Hamilton General or Juravinski Hospitals following a fall are eligible for recruitment
Sampling Method: Non-Probability Sample
Enrollment: 1753 (Actual)
Dates: Start 2015-12-14 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Intracranial Bleeding | 6 weeks
  the incidence of intracranial bleeding (including subdural, subarachnoid, extradural, intracerebral and cerebral contusion) diagnosis in the following 6 weeks

SECONDARY OUTCOMES:
Proportion of immediate bleeds | 6 weeks
  Intracranial bleeding categorized as 'immediate' and 'delayed', neurosurgical intervention for intracranial bleeding, length of stay in hospital and all cause mortality at 6 weeks.
Proportion of delayed bleeds | 6 weeks
  Intracranial bleeding categorized as 'immediate' and 'delayed', neurosurgical intervention for intracranial bleeding, length of stay in hospital and all cause mortality at 6 weeks.
Proportion Eligible | Duration of Recruitment
  Proportion of eligible patients identified, recruited and followed up

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin de Wit, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton Health Ciences, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No